CLINICAL TRIAL: NCT03221504
Title: 7-day Compared With 10-day Antibiotic Treatment for Febrile Urinary Tract Infections in Children: a Randomized Controlled Trial
Brief Title: 7-day Compared With 10-day Antibiotic Treatment for Febrile Urinary Tract Infections in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WUM
Record Dates: First submitted 2017-07-07; First posted 2017-07-18 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2017-07

CONDITIONS: Urinary Tract Infections in Children
Keywords: urinary tract infections; pyelonephritis; cefuroxime; children
MeSH Terms: conditions — Urinary Tract Infections; Pyelonephritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antibiotic therapy for 10 days (Active Comparator): After 7 days of cefuroxime treatment (oral, intravenous or sequential), patients from day 8 to day 10 will continue to receive the antibiotic (in blinded bottle).
  Interventions: Other: Longer therapy duration
- Antibiotic therapy for 7 days (Experimental): After 7 days of cefuroxime therapy (oral, intravenous or sequential), children from day 8 to day 10 will receive placebo (in blinded bottle).
  Interventions: Other: Shorter therapy duration

INTERVENTIONS:
Other: Longer therapy duration — Patients will receive cefuroxime axetil orally. Treatment will involve the supply of cefuroxime axetil 30 mg/kg/d in two divided doses (in blinded bottles).
  Arms: Antibiotic therapy for 10 days
Other: Shorter therapy duration — Patients will receive placebo orally (in blinded bottles). The volume of the placebo will be like cefuroxime syrup.
  Arms: Antibiotic therapy for 7 days

SUMMARY:
The investigators aim to assess the effectiveness of a 7-day compared with a 10-day course of antibiotic treatment for febrile urinary tract infections (UTIs) in children. It is formulated a hypothesis that a 7-day course of antibiotic therapy is equally effective as a 10-day course of therapy and would entail a lower risk of adverse events and better compliance.

DETAILED DESCRIPTION:
In previously published European and global guidelines, there has been no consensus among experts regarding the duration of therapy for a febrile UTI. Depending on the recommendation, the duration of treatment should be between 7-14 days.

221 patients aged 3 months to 7 years with febrile UTIs (defined as a combination of fever and leukocyturia in urine sediment) will be randomly assigned to receive a 7-day treatment arm (7 days of cefuroxime/cefuroxime axetil followed by 3 days of blinded placebo) or a 10-day treatment arm (7 days of cefuroxime/cefuroxime axetil followed by 3 days of blinded cefuroxime axetil).

The primary outcome measure will be frequencies of recurrence and reinfection of UTI during the 6 months after the intervention. The secondary outcome measures will be antibiotic-associated diarrhea and compliance.

ELIGIBILITY:
Inclusion Criteria (must have all):

* children aged from 3 months to 7 years
* clinical diagnosis of a febrile UTI at presentation according to urinalysis (white blood cells in the sediment >10 in the field of view);
* fever ≥38°C
* positive urine collection with sensitivity for cefuroxime
* treatment cefuroxime or cefuroxime axetil for 7 days

Exclusion Criteria (must have one):

* history of a UTI in the last 3 months
* prophylaxis for UTI
* antibiotic therapy in the last month
* known allergy to the study drugs
* immunosuppression therapy
* disease with immune deficiency
* children with other coexisting infection, e.g. meningitis, sepsis, pneumonia, otitis
* severe obstructive uropathy

Ages: 3 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 221 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
frequencies of recurrence of UTI | 3 months after intervention
  New onset of symptomatic UTI within the 3 months follow-up period. The recurrence of a UTI is diagnosed when the next infection is caused by the same microorganism during 3 months following the treatment of a UTI.

SECONDARY OUTCOMES:
frequencies of reinfection of UTI | 6 months after intervention
  The reinfection of a UTI is diagnosed when the next infection is caused by a different bacteria.
antibiotic-associated diarrhoea (AAD), compliance | 7 days after intervention
  AAD is defined by the daily production of at least 3 loose or watery stools for at least 48 hours during antibiotic treatment and 7 days after administration of the antibiotic.
  Compliance with the study protocol will be assessed by direct interview with the patient and/or caregiver and by measuring the amount of the fluid left in the bottle at the end of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Pańczyk-Tomaszewska, Assistant Professor, Study Chair — Medical Univeristy of Warsaw; Maria Daniel, MD, Principal Investigator — Medical Univeristy of Warsaw
Locations (2):
- Poland (2):
  - Children's Hospital for The Medical University of Warsaw, Warsaw
  - The Holy Family Specialistic Hospital, Warsaw

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Simoes e Silva AC, Oliveira EA. Update on the approach of urinary tract infection in childhood. J Pediatr (Rio J). 2015 Nov-Dec;91(6 Suppl 1):S2-10. doi: 10.1016/j.jped.2015.05.003. Epub 2015 Sep 7. PMID 26361319
- [Background] Conway PH, Cnaan A, Zaoutis T, Henry BV, Grundmeier RW, Keren R. Recurrent urinary tract infections in children: risk factors and association with prophylactic antimicrobials. JAMA. 2007 Jul 11;298(2):179-86. doi: 10.1001/jama.298.2.179. PMID 17622599
- [Background] Craig JC, Simpson JM, Williams GJ, Lowe A, Reynolds GJ, McTaggart SJ, Hodson EM, Carapetis JR, Cranswick NE, Smith G, Irwig LM, Caldwell PH, Hamilton S, Roy LP; Prevention of Recurrent Urinary Tract Infection in Children with Vesicoureteric Reflux and Normal Renal Tracts (PRIVENT) Investigators. Antibiotic prophylaxis and recurrent urinary tract infection in children. N Engl J Med. 2009 Oct 29;361(18):1748-59. doi: 10.1056/NEJMoa0902295. PMID 19864673
- [Background] Subcommittee on Urinary Tract Infection, Steering Committee on Quality Improvement and Management; Roberts KB. Urinary tract infection: clinical practice guideline for the diagnosis and management of the initial UTI in febrile infants and children 2 to 24 months. Pediatrics. 2011 Sep;128(3):595-610. doi: 10.1542/peds.2011-1330. Epub 2011 Aug 28. PMID 21873693
- [Background] Montini G, Toffolo A, Zucchetta P, Dall'Amico R, Gobber D, Calderan A, Maschio F, Pavanello L, Molinari PP, Scorrano D, Zanchetta S, Cassar W, Brisotto P, Corsini A, Sartori S, Da Dalt L, Murer L, Zacchello G. Antibiotic treatment for pyelonephritis in children: multicentre randomised controlled non-inferiority trial. BMJ. 2007 Aug 25;335(7616):386. doi: 10.1136/bmj.39244.692442.55. Epub 2007 Jul 4. PMID 17611232
- [Background] Michael M, Hodson EM, Craig JC, Martin S, Moyer VA. Short versus standard duration oral antibiotic therapy for acute urinary tract infection in children. Cochrane Database Syst Rev. 2003;(1):CD003966. doi: 10.1002/14651858.CD003966. PMID 12535494
- [Background] Ammenti A, Cataldi L, Chimenz R, Fanos V, La Manna A, Marra G, Materassi M, Pecile P, Pennesi M, Pisanello L, Sica F, Toffolo A, Montini G; Italian Society of Pediatric Nephrology. Febrile urinary tract infections in young children: recommendations for the diagnosis, treatment and follow-up. Acta Paediatr. 2012 May;101(5):451-7. doi: 10.1111/j.1651-2227.2011.02549.x. Epub 2012 Jan 3. PMID 22122295
- [Derived] Daniel M, Szajewska H, Panczyk-Tomaszewska M. 7-day compared with 10-day antibiotic treatment for febrile urinary tract infections in children: protocol of a randomised controlled trial. BMJ Open. 2018 Mar 2;8(3):e019479. doi: 10.1136/bmjopen-2017-019479. PMID 29500209
- See also: National Institute for Health and Care Excellence. Urinary tract infections in children and young people 2013 July — https://www.nice.org.uk/guidance/qs36
- See also: European Association of Urology; European Society for Pediatric Urology Urinary tract infections in children: EAU/ESPU guidelines. — http://uroweb.org/guideline/paediatric-urology/#3
- See also: Canadian Paediatric Society, Urinary tract infection in infants and children: Diagnosis and management — http://www.cps.ca/en/documents/position/urinary-tract-infections-in-children